CLINICAL TRIAL: NCT05926544
Title: Addressing COVID-19 Vaccine Hesitancy in Rural Community Pharmacies Reducing Disparities Through an Implementation Science Approach
Brief Title: COVID-19 Vaccine Hesitancy Counseling Intervention for Pharmacists
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not receiving primary outcome data needed
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Arkansas (Other); University of South Carolina (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 22-2602a; 1R01MD018085 (NIH)
Record Dates: First submitted 2023-06-28; First posted 2023-07-03 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-03

CONDITIONS: COVID-19
Keywords: vaccine hesitancy; fidelity; vaccination
MeSH Terms: conditions — COVID-19; Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: The investigators will use an incomplete stepped wedge cluster randomized design, where units (pharmacies) begin in one condition (standard implementation approach) and "crossover" to the other condition (virtual facilitation).
Who Masked: Outcomes Assessor
Masking Description: Study staff who are rating fidelity will be blinded to whether the observation is from the standard implementation or virtual facilitation condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard implementation (Stage 1) (Experimental): Participants begin with the standard implementation interventions for 8-16 weeks, depending on random block assignment.
  Interventions: Behavioral: Standard implementation webinar and online training
- Virtual facilitation (Stage 2) (Experimental): After completing the standard implementation, participants then complete the virtual facilitation intervention for 8-16 weeks, depending on random block assignment.
  Interventions: Behavioral: Virtual facilitation

INTERVENTIONS:
Behavioral: Standard implementation webinar and online training — The one-hour webinar (either live or pre-recorded) will include updated information about the COVID-19 virus, variant nomenclature, booster eligibility, mechanisms of action, and outcomes.
  The 30-minute online training addresses how to communicate about COVID-19 vaccinations, presents a 5-step process for initiating conversations, includes example verbiage about how to address specific concerns, and has example videos that show how to implement the 5-step process with vaccine hesitant patients.
  Arms: Standard implementation (Stage 1)
Behavioral: Virtual facilitation — This intervention involves a 30-minute virtual facilitation site visit and 8 30-minute virtual facilitator coaching sessions. The virtual site visit over Zoom will establish the personnel and workflows at each pharmacy and allow the facilitator to establish rapport. Weekly Zoom calls will allow the virtual facilitator to work with a participant to review overall implementation challenges associated with approaching patients, delivering the intervention, and documenting results. Lastly, either the facilitator or the participant can request and schedule a Zoom call to go over any pressing implementation issue in need of rapid attention (e.g., technical difficulties with the website).
  Arms: Virtual facilitation (Stage 2)

SUMMARY:
The goal of this clinical trial is to test if virtual facilitation (e.g., video coaching) increases rural pharmacists' ability to implement COVID-19 vaccine hesitancy counseling when compared to a "standard" implementation approach (e.g., training and dissemination of implementation support tools) in rural pharmacies. The main question it aims to answer is if virtual facilitation improves fidelity to a newly developed vaccine hesitancy counseling intervention when compared to standard implementation.

All participants will begin in the standard implementation condition, where they will complete a webinar on COVID-19 vaccinations and a 30-minute online training on vaccine hesitancy communication. After standard implementation, they will switch to the virtual facilitation condition where they will be assigned a virtual coach to help them with implementing the intervention. There will be four fidelity observations per each 8-week intervention period to determine whether pharmacists are implementing the intervention as intended. Researchers will compare fidelity between the standard and virtual facilitation conditions.

DETAILED DESCRIPTION:
Because COVID-19 vaccination conversations are sensitive and often politically charged, pharmacists need implementation support, including training and ongoing guidance to deliver evidence-based vaccine hesitancy counseling interventions. Implementation facilitation, in which trained facilitators coach and troubleshoot problems with professionals as they implement new practices, increases adoption of practices with fidelity. However, implementation facilitation generally, and virtual facilitation (e.g., video coaching) in particular, has not been systematically studied in community pharmacy settings.

The goal of this study is to test if virtual facilitation increases rural pharmacists' ability to implement COVID-19 vaccine hesitancy counseling when compared to a "standard" implementation approach (e.g., training and dissemination of implementation support tools). Using a rural pharmacy practice-based research network (PBRN) that spans 7 southeastern states, the investigators will conduct a stepped-wedge trial with 30 rural pharmacies to test whether virtual facilitation outperforms the standard approach in increasing the fidelity with which pharmacists implement the vaccine hesitancy counseling intervention. Using a project-sponsored data collection system, the investigators will gather data on implementation outcomes, including fidelity and effectiveness.

All participants will begin in the standard implementation condition, where they will complete a webinar on COVID-19 vaccinations and a 30-minute online training on vaccine hesitancy communication. After the standard implementation period, they will crossover to the virtual facilitation condition where they will be assigned a virtual coach to help them with implementing the intervention. There will be four fidelity observations per each 8-week intervention period to determine whether pharmacists are implementing the intervention as intended. Researchers will compare fidelity between the standard and virtual facilitation conditions. Based on a proposed Fall 2023 vaccine administration schedule by the Federal Drug Administration, we anticipate implementing the study over two vaccination seasons (Fall 2023 and Fall 2024).

ELIGIBILITY:
Inclusion Criteria:

* The pharmacy must be a member of the Rural Research Alliance for Community Pharmacies (RURAL-CP)
* The pharmacy must be located in a county that has an African American population of at least 32.9% or had at least 58% of the population vote for a Republican president in 2020.

Exclusion Criteria:

* The pharmacy will be excluded if it does not offer COVID-19 primary series or booster vaccines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Delesha M Carpenter, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Geoffrey Curran, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Curran GM, Shoemaker SJ. Advancing pharmacy practice through implementation science. Res Social Adm Pharm. 2017 Sep-Oct;13(5):889-891. doi: 10.1016/j.sapharm.2017.05.018. Epub 2017 Jun 1. No abstract available. PMID 28619650
- [Background] Bauer MS, Miller CJ, Kim B, Lew R, Stolzmann K, Sullivan J, Riendeau R, Pitcock J, Williamson A, Connolly S, Elwy AR, Weaver K. Effectiveness of Implementing a Collaborative Chronic Care Model for Clinician Teams on Patient Outcomes and Health Status in Mental Health: A Randomized Clinical Trial. JAMA Netw Open. 2019 Mar 1;2(3):e190230. doi: 10.1001/jamanetworkopen.2019.0230. PMID 30821830
- [Background] Curran GM, Mukherjee S, Allee E, Owen RR. A process for developing an implementation intervention: QUERI Series. Implement Sci. 2008 Mar 19;3:17. doi: 10.1186/1748-5908-3-17. PMID 18353186
- [Background] Knox L. Module 2: Practice Facilitation as a Resource for Practice Improvement. In: Quality AfHRa, ed. pcmh.ahrq.gov: AHRQ; 2015.
- [Background] Parchman ML, Noel PH, Culler SD, Lanham HJ, Leykum LK, Romero RL, Palmer RF. A randomized trial of practice facilitation to improve the delivery of chronic illness care in primary care: initial and sustained effects. Implement Sci. 2013 Aug 22;8:93. doi: 10.1186/1748-5908-8-93. PMID 23965255
- [Derived] Curran G, Mosley C, Gamble A, Painter J, Ounpraseuth S, Brewer NT, Teeter B, Smith M, Halladay J, Hughes T, Shepherd JG, Hastings T, Simpson K, Carpenter D. Addressing COVID-19 vaccine hesitancy in rural community pharmacies: a protocol for a stepped wedge randomized clinical trial. Implement Sci. 2023 Dec 18;18(1):72. doi: 10.1186/s13012-023-01327-7. PMID 38110979

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Pharmacies begin with the standard implementation interventions for 8-16 weeks and after completing the standard implementation, then complete the virtual facilitation intervention for 8-16 weeks, then move into follow-up period for 8 weeks.
Units Other Than Participants: Pharmacy
Groups:
- Sequence 1: Oct-Nov 23 8 Weeks Standard, Dec-Jan 8 Weeks Facilitation, Feb-Mar 24 8 Weeks Follow Up: Pharmacies begin with the standard implementation intervention for 8 weeks. This involves a webinar and online training. The 1-hour webinar (either live or pre-recorded) includes updated information about the COVID-19 virus, variant nomenclature, booster eligibility, mechanisms of action, and outcomes. The 30-minute online training addresses how to communicate about COVID-19 vaccinations, presents a 5-step process for initiating conversations, includes example verbiage about how to address specific concerns, and has example videos that show how to implement the 5-step process with vaccine hesitant patients.
  After completing the standard implementation, pharmacies then complete the virtual facilitation intervention for 8 weeks. This involves a 30-minute virtual facilitation site visit and 8 30-minute virtual facilitator coaching sessions. The virtual site visit over Zoom establishes the personnel and workflows at each pharmacy and allows the facilitator to establish rapport. Weekly Zoom calls allow the virtual facilitator to work with a pharmacy to review overall implementation challenges associated with approaching patients, delivering the intervention, and documenting results. After completing the virtual facilitation, pharmacies move into follow-up period for 8 weeks.
- Sequence 2: Oct 23-Jan 24 16 Weeks Standard, Feb-Mar 8 Weeks Facilitation, Aug-Sep 8 Weeks Follow up: Pharmacies begin with the standard implementation intervention for 16 weeks. This involves a webinar and online training. The 1-hour webinar (either live or pre-recorded) includes updated information about the COVID-19 virus, variant nomenclature, booster eligibility, mechanisms of action, and outcomes. The 30-minute online training addresses how to communicate about COVID-19 vaccinations, presents a 5-step process for initiating conversations, includes example verbiage about how to address specific concerns, and has example videos that show how to implement the 5-step process with vaccine hesitant patients.
  After completing the standard implementation, pharmacies then complete the virtual facilitation intervention for 8 weeks. This involves a 30-minute virtual facilitation site visit and 8 30-minute virtual facilitator coaching sessions. The virtual site visit over Zoom establishes the personnel and workflows at each pharmacy and allows the facilitator to establish rapport. Weekly Zoom calls allow the virtual facilitator to work with a pharmacy to review overall implementation challenges associated with approaching patients, delivering the intervention, and documenting results. After completing the virtual facilitation, pharmacies move into follow-up period for 8 weeks.
- Sequence 3: Oct-Nov 23 8 Weeks Standard, Dec-Mar 16 Weeks Facilitation, Aug-Sep 24 8 Weeks Follow up: Pharmacies begin with the standard implementation intervention for 8 weeks. This involves a webinar and online training. The 1-hour webinar (either live or pre-recorded) includes updated information about the COVID-19 virus, variant nomenclature, booster eligibility, mechanisms of action, and outcomes. The 30-minute online training addresses how to communicate about COVID-19 vaccinations, presents a 5-step process for initiating conversations, includes example verbiage about how to address specific concerns, and has example videos that show how to implement the 5-step process with vaccine hesitant patients.
  After completing the standard implementation, pharmacies then complete the virtual facilitation intervention for 16 weeks. This involves a 30-minute virtual facilitation site visit and 8 30-minute virtual facilitator coaching sessions. The virtual site visit over Zoom establishes the personnel and workflows at each pharmacy and allows the facilitator to establish rapport. Weekly Zoom calls allow the virtual facilitator to work with a pharmacy to review overall implementation challenges associated with approaching patients, delivering the intervention, and documenting results. After completing the virtual facilitation, pharmacies move into follow-up period for 8 weeks.
Period: Oct-Nov 2023
Arm/Group | Sequence 1: Oct-Nov 23 8 Weeks Standard, Dec-Jan 8 Weeks Facilitation, Feb-Mar 24 8 Weeks Follow Up | Sequence 2: Oct 23-Jan 24 16 Weeks Standard, Feb-Mar 8 Weeks Facilitation, Aug-Sep 8 Weeks Follow up | Sequence 3: Oct-Nov 23 8 Weeks Standard, Dec-Mar 16 Weeks Facilitation, Aug-Sep 24 8 Weeks Follow up
Started | 6; 6 Pharmacy | 5; 5 Pharmacy | 5; 5 Pharmacy
Completed | 5; 5 Pharmacy | 5; 5 Pharmacy | 5; 5 Pharmacy
Not Completed | 1; 1 Pharmacy | 0; 0 Pharmacy | 0; 0 Pharmacy
Period: Dec 2023-Jan 2024
Arm/Group | Sequence 1: Oct-Nov 23 8 Weeks Standard, Dec-Jan 8 Weeks Facilitation, Feb-Mar 24 8 Weeks Follow Up | Sequence 2: Oct 23-Jan 24 16 Weeks Standard, Feb-Mar 8 Weeks Facilitation, Aug-Sep 8 Weeks Follow up | Sequence 3: Oct-Nov 23 8 Weeks Standard, Dec-Mar 16 Weeks Facilitation, Aug-Sep 24 8 Weeks Follow up
Started | 5; 5 Pharmacy | 5; 5 Pharmacy | 5; 5 Pharmacy
Completed | 5; 5 Pharmacy | 4; 4 Pharmacy | 5; 5 Pharmacy
Not Completed | 0; 0 Pharmacy | 1; 1 Pharmacy | 0; 0 Pharmacy
Period: Feb-Mar 2024
Arm/Group | Sequence 1: Oct-Nov 23 8 Weeks Standard, Dec-Jan 8 Weeks Facilitation, Feb-Mar 24 8 Weeks Follow Up | Sequence 2: Oct 23-Jan 24 16 Weeks Standard, Feb-Mar 8 Weeks Facilitation, Aug-Sep 8 Weeks Follow up | Sequence 3: Oct-Nov 23 8 Weeks Standard, Dec-Mar 16 Weeks Facilitation, Aug-Sep 24 8 Weeks Follow up
Started | 5; 5 Pharmacy | 4; 4 Pharmacy | 5; 5 Pharmacy
Completed | 1; 1 Pharmacy | 4; 4 Pharmacy | 5; 5 Pharmacy
Not Completed | 4; 4 Pharmacy | 0; 0 Pharmacy | 0; 0 Pharmacy
Period: Aug-Sep 2024
Arm/Group | Sequence 1: Oct-Nov 23 8 Weeks Standard, Dec-Jan 8 Weeks Facilitation, Feb-Mar 24 8 Weeks Follow Up | Sequence 2: Oct 23-Jan 24 16 Weeks Standard, Feb-Mar 8 Weeks Facilitation, Aug-Sep 8 Weeks Follow up | Sequence 3: Oct-Nov 23 8 Weeks Standard, Dec-Mar 16 Weeks Facilitation, Aug-Sep 24 8 Weeks Follow up
Started | 0; 0 Pharmacy (Not applicable for participants in Sequence 1. These participants were not assigned to any study activities for Aug-Sep 2024.) | 0; 0 Pharmacy (Follow-up not completed due to study termination.) | 0; 0 Pharmacy (Follow-up not completed due to study termination.)
Completed | 0; 0 Pharmacy | 0; 0 Pharmacy | 0; 0 Pharmacy
Not Completed | 0; 0 Pharmacy | 0; 0 Pharmacy | 0; 0 Pharmacy

BASELINE CHARACTERISTICS:
Population: The unit of analysis is pharmacy and no baseline characteristics were collected.
Units Other Than Participants: Pharmacy
Groups:
- Block 1 Standard Implementation; Block 2 Standard Implementation; Block 3 Standard Implementation: Pharmacies begin with the standard implementation interventions for 8-16 weeks.
- Total: Total of all reporting groups
Arm/Group | Block 1 Standard Implementation | Block 2 Standard Implementation | Block 3 Standard Implementation | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Number analyzed (Pharmacy) | 0 | 0 | 0 | 0
Age, Categorical — Population: Age data were not collected.
Sex: Female, Male — Population: Sex data were not collected.
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean Fidelity Score
Description: The fidelity measure focuses on the competence and skill of the pharmacist (7 items with values ranging from 1 to 3) in their delivery of the vaccine hesitancy counseling intervention. Items assess whether they expressed empathy, used non-confrontational manner, spoke confidently without using jargon, emphasized patient autonomy, reflected back patient's statements accurately, and used a respectful demeanor. The overall composite competency score is the sum of the 7 items with scores ranging from 7 to 21, with higher scores reflecting greater competency in the delivery of the vaccine hesitancy intervention. Fidelity will be measured for each pharmacist four times per each 8-week intervention period under the standard implementation approach and the virtual facilitation approach. In pharmacies with more than one pharmacist, fidelity ratings will be averaged to achieve a pharmacy-level measure.
Time Frame: From baseline through the end of the virtual facilitation periods, up to 24 weeks max.
Population: Pharmacists were unable to record actual conversations at the pharmacy and the approach was changed to a standardized patient audio recording. This change was made towards the end of the Standard implementation period thus only 1 pharmacy provided data using the viable method. Data successfully collected from 9 pharmacies in the Virtual facilitation period.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Pharmacies
Groups:
- Standard Implementation (Stage 1): Pharmacies begin with the standard implementation interventions for 8-16 weeks, depending on random block assignment.
  Standard implementation webinar and online training: The one-hour webinar (either live or pre-recorded) will include updated information about the COVID-19 virus, variant nomenclature, booster eligibility, mechanisms of action, and outcomes.
  The 30-minute online training addresses how to communicate about COVID-19 vaccinations, presents a 5-step process for initiating conversations, includes example verbiage about how to address specific concerns, and has example videos that show how to implement the 5-step process with vaccine hesitant patients.
- Virtual Facilitation (Stage 2): After completing the standard implementation, participants then complete the virtual facilitation intervention for 8-16 weeks, depending on random block assignment.
  Virtual facilitation: This intervention involves a 30-minute virtual facilitation site visit and 8 30-minute virtual facilitator coaching sessions. The virtual site visit over Zoom will establish the personnel and workflows at each pharmacy and allow the facilitator to establish rapport. Weekly Zoom calls will allow the virtual facilitator to work with a pharmacy to review overall implementation challenges associated with approaching patients, delivering the intervention, and documenting results. Lastly, either the facilitator or the participant can request and schedule a Zoom call to go over any pressing implementation issue in need of rapid attention (e.g., technical difficulties with the website).
Arm/Group | Standard Implementation (Stage 1) | Virtual Facilitation (Stage 2)
Number analyzed (Participants) | 1 | 9
Number analyzed (Pharmacies) | 1 | 9
score on a scale | 20 (0) | 15.82 (2.06)

2. Secondary Outcome: Proportion of Individuals Receiving Vaccine Hesitancy Counseling Who Chose to Get the COVID-19 Vaccine
Description: Effectiveness will be calculated as the proportion of patients who received the vaccine hesitancy counseling intervention who chose to get the COVID-19 vaccine. Pharmacists at each pharmacy were asked to document 30 conversations (10 per 8-week period). Pharmacists documented whether each of the patients elected to get the COVID-19 vaccine after their conversation.
Time Frame: From baseline through the end of the virtual facilitation periods, up to 24 weeks maximum
Population: Not all pharmacists documented their conversations with COVID vaccine hesitant patients, resulting in missing data from both the standard implementation and virtual facilitation periods.
Measure: Number; unit: Proportion of patients vaccinated
Units Other Than Participants: Conversations documented
Arm/Group | Standard Implementation (Stage 1) | Virtual Facilitation (Stage 2)
Number analyzed (Participants) | 11 | 9
Number analyzed (Conversations documented) | 85 | 82
Proportion of patients vaccinated | 0.38 | 0.20
Statistical Analysis 1: Comparison: Standard Implementation (Stage 1) vs Virtual Facilitation (Stage 2); Test type: Superiority; Risk Ratio (RR) = 0.46, 95% CI 2-sided [0.18 to 1.16] — The Standard implementation arm was the reference group

ADVERSE EVENTS:
Time Frame: This study did not monitor for untoward medical occurrences/adverse events.
Description: Per the study protocol, participating pharmacists were not considered to be at risk for medically-related adverse events. An example of a relevant "adverse event" would be a data breach which although study-related is not a medical event. Therefore, adverse events data collection was not a part of this protocol.
Groups:
- Block 1 Standard Implementation; Block 2 Standard Implementation; Block 3 Standard Implementation: Participants begin with the standard implementation interventions for 8-16 weeks.
  Standard implementation webinar and online training: The one-hour webinar (either live or pre-recorded) will include updated information about the COVID-19 virus, variant nomenclature, booster eligibility, mechanisms of action, and outcomes.
  The 30-minute online training addresses how to communicate about COVID-19 vaccinations, presents a 5-step process for initiating conversations, includes example verbiage about how to address specific concerns, and has example videos that show how to implement the 5-step process with vaccine hesitant patients.
- Block 1 Virtual Facilitation; Block 2 Virtual Facilitation; Block 3 Virtual Facilitation: After completing the standard implementation, participants then complete the virtual facilitation intervention for 8-16 weeks.
  Virtual facilitation: This intervention involves a 30-minute virtual facilitation site visit and 8 30-minute virtual facilitator coaching sessions. The virtual site visit over Zoom will establish the personnel and workflows at each pharmacy and allow the facilitator to establish rapport. Weekly Zoom calls will allow the virtual facilitator to work with a participant to review overall implementation challenges associated with approaching patients, delivering the intervention, and documenting results. Lastly, either the facilitator or the participant can request and schedule a Zoom call to go over any pressing implementation issue in need of rapid attention (e.g., technical difficulties with the website).
- Block 1 Follow-Up; Block 2 Follow-Up; Block 3 Follow-Up: After completing the virtual facilitation, participants move into follow-up period for 8 weeks.
Arm/Group | Block 1 Standard Implementation | Block 1 Virtual Facilitation | Block 1 Follow-Up | Block 2 Standard Implementation | Block 2 Virtual Facilitation | Block 2 Follow-Up | Block 3 Standard Implementation | Block 3 Virtual Facilitation | Block 3 Follow-Up
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-19): https://cdn.clinicaltrials.gov/large-docs/44/NCT05926544/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT05926544/ICF_000.pdf